CLINICAL TRIAL: NCT05192447
Title: Analysis of the Cognitive-behavioral Dysfunctions Profile and the Potential of Neuroplasticity in Patients With Brain Tumors Subjected to Selected Radiotherapy Techniques and the Possibility of Their Compensation by Psycho-physical Training
Brief Title: The Cognitive-Behavioral Dysfunctions and the Potential of Neuroplasticity in Brain Tumors Patients During Radiotherapy
Acronym: REHABrain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Greater Poland Cancer Centre (Other)
Collaborators: National Science Centre, Poland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2020/37/B/NZ7/01122; 480821 (Registry Identifier: National Science Centre Poland)
Record Dates: First submitted 2021-06-29; First posted 2022-01-14 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Brain Tumors; Radiotherapy
Keywords: neuroplasticity; rehabilitation
MeSH Terms: conditions — Brain Neoplasms | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group = Exercise Group (Experimental): EG will perform complementary cognitive and physical training (120 min./5/per week during study observation)
  Interventions: Behavioral: Exercise treatment
- Control Group (No Intervention): CG will be provided with normal hospital care during RT and next will conduct a normal daily activity at home.

INTERVENTIONS:
Behavioral: Exercise treatment — Patients selected to EG will carry out complementary cognitive and physical training under supervision of rehabilitation staff. For neuropsychological exercises, the investigators will use the RehaCom system - high quality scientific neurocognitive disorder therapy programs and software. (Time: 30 min./5 times/week per patient during RT). In this time, EG patients will do physical training (such as cycling, running on properly calibrated equipment for the circulatory system parameter measurement (1hour/ 5 days/ week), and neuromuscular and cognitive reeducation exercises using a technically advanced tool - Neuroforma computer software - 30 min/ 5 times/ week). After the end of RT, patients in EG will do a special exercise training at home under supervision of staff from the Department of Rehabilitation, and cognitive training using special tasks (3 times an hour/per week) at home, and two times/week using RehaCom and Neuroforma (60 min/sesion) in our cancer ceter.
  Other Names: Rehabilitation treatment
  Arms: Intervention Group = Exercise Group

SUMMARY:
Primary and secondary brain tumors are a constant challenge for the medicine. Tissue sensitivity to ionizing radiation differs and depends on numerous factors and the same dose of radiation may produce different effects in particular structures of the CNS. It can also affect the surrounding healthy tissues and lead to adverse effects like the cognitive or physical function impairment. One of brain structures most sensitive to ionizing radiation is the limbic system, especially the hippocampus, because it is here that the postnatal neurogenesis takes place via neural stem cells, which are a self-renewing population of precursor cells. There have been no studies that would thoroughly examine the impact of different CNS radiation therapy techniques on the cognitive function, potential neuroplasticity markers or blood-brain barrier damage in brain tumor patients with a concomitant use of neurocognitive combination therapies or physical exercise, and their impact on the CNS function.

The aim of the study is to assess the impact of selected RT techniques: IMRT, WBRT, and CyberKnife (SRS) on the processes regulating cognitive and physical function in patients with primary (Group III and IV, WHO, 2016) and metastatic CNS tumors. The secondary objective is the analysis of the effect of selected forms of neurorehabilitation on the parameters studied. The study will be a prospective clinical trial conducted in 150 patients. Patient evaluation will be carried out before RT, after RT, during a follow-up visit-3 months after RT, and finally after 6 months. The methods will be used: analysis of the blood-brain barrier permeability markers including exact connection proteins, markers confirming neuroplasticity of the brain, cerebral secretory activity, and onco- and anti-neuronal antibody activity, brain structure analysis (MRI) and volume testing of selected brain structures, and assessment of cognitive and physical function of the patients. The study will be a part of the search trend aiming to explain the mechanism of the formation of cognitive-behavioral disorders in humans based on the most fundamental principles governing information processing in CNS, and the impact of neoplasia and ionizing radiation on selected brain structures and functions. The results of the study might become a starting point for the formulation of new guidelines on the level of physical activity or cognitive exercise in patients treated with CNS radiation therapy.

DETAILED DESCRIPTION:
Every year, thousands of patients worldwide undergo radiotherapy (RT) for primary brain tumors (BT) and brain metastases originating from extracranial tumors. Radiation injury is multifactorial and is characterized by e.g. vascular abnormalities, inflammation, gliosis, demyelination, and often at high doses, white matter necrosis. Standard treatment of BT includes high dose megavoltage radiation to the cranial vault, but 50-90% of overall survivors exhibit impaired cognition and functional dysfunction. The radiation cognitive syndrome is still poorly understood, and there is no effective prevention or long-term treatment. Therefore, the investigators will analyze specific molecular markers which may have a relationship with morfological changes in the brain, its secretive and imunological role as well as cognitive function and postulate that previously undetected and comparatively subtle early manifestations of irradiation damage to CNS may synergize over time to form macro- and microstructural abnormalities. The investigators plan to corroborate a hypothesis that impairment of cognitive and motor functions in patients undergoing RT can be limited. In study, the investigators will quantitatively and objectively evaluate the effects of exercise on brain activity during cognitive and physical training in BT patients treated with RT. Therefore, specific objectives include: 1. Analysis of the molecular mechanism in BBB disruption. 2. Multidimensional analysis of specific neuroplasticity markers, onconeural-antibodies etc. 3. Assessment of the volume of the brain structures and their morphology. 4. Analysis of the results of neurocognitive and functional tests.

Significance of the project The Response Assessment in Neuro-Oncology working group recommended that neurocognitive outcome should be considered one of the primary endpoints in BT clinical trials. Despite the importance and clear concern about radiation-induced cognitive decline, the pathophysiology driving the progression of this syndrome remains poorly understood, and there are no effective preventative measures or long-term treatments. To date, there has been no study comparing different techniques of irradiation, namely intensity-modulated photon RT (IMRT), whole brain RT (WBRT), and stereotactic radiosurgery (CyberKnife), in BT patients in the aspect of pathophysiology of BBB or immunological aspects, as well as neurogenesis, neuroplasticity. These methods will be rely on a detailed understanding of radiation dose-volume effects, which link the incidence and severity of neurocognitive and functional impairment to specific volumes and morphology of normal brain. Possible explanations for the preservation of cognition and behavior include the resiliency of the cerebellum, frontal and tempo-parietal lobes, the hippocampus-mammillary complex and other supratentorial regions. Radiation is now known to suppress the proliferation of progenitor cells and their differentiation into neurons. The relatively recent discovery of neural stem cells in discrete areas of the brain is the impetus behind the most recent potential target for radiation. Early changes below the gross anatomical level, including a decline in neurogenesis, microvascular damage, subtle loss of white matter integrity, and disturbances of neuronal morphophysiology, may interact and progressively alter neuronal stem cell niches to impede neuronal function, viability, and progenitor cell differentiation. Therefore, the investigators will thoroughly observe the mechanism of neurogenesis and the possible improvement of neuroprotection and neuroregeneration in BT patients undergoing various forms of RT. Previous research has shown that physical exercise in healthy people is associated with increased structural and functional integrity in regions that overlap with brain functions, including the frontal, motor cortex, and the cerebellum. The precise neurobiological mechanism for cognitive effects of rehabilitation remains unknown, however a vast rodent literature supports a central role of protective neurotrophins, which have been shown to facilitate production of new neurons in the hippocampus, promote synaptic plasticity in cerebral cortex, and enhance growth and protection of neurovasculature and suggests exercise may promote formation and strengthening of connections between the hippocampus and its widespread cortical connections, which improve cognitive and behaviour functioning. However, the specific brain structure and function regions activated during rehabilitation exercise in patients with BT during oncological treatment still remain largely undefined. The study results obtained in this project will provide new knowledge about metabolic and structural pathways of the CNS in the context of RT and will also provide the basis for the development of regenerative medicine in oncology.

Work plan The investigators will conduct study in the Greater Poland Cancer Centre. The participants will be enrolled in this study according study criteria from the Department of Radiotherapy after medical assessment by an oncologist (physician). Evaluation of the all subjects will be carried out: at baseline (T0), one month after RT (T1), and control (T2) - 3 months after RT and final (T3) - 6 months after RT (unless there is a deterioration of health making the assessment impossible, or death). The investigators will monitor the patients by:

A. Analysis of the patient's blood serum: 1/ markers of BBB disruption: S-100β and circulating tight junction-related proteins (occludin, claudin-5, zonula occludens-1); 2/ factors with potential effect on neuroplasticity - immune-cell production of neurotrophins e.g. brain-derived neurotrophic factor, beta-nerve growth factor, neurotrophin-3, neurotrophin-4/5; 3/ activity of carnosinase and its isoenzymes; 4/ onconeural antibodies (anti-Hu, anti-Ri, anti-Yo, anti-Ma/Ta, anti-Cv2, and anti-amphiphysin as well as anti-myelin, anti-MAG, anti-GAD) and anti-surface neuronal antigens (anti-NMDA, anti-AMPA, anti-GABA, anti-DPPX, anti-LGI1, anti-CASPR) to investigate correlations with types of BT, RT, and possible paraneoplastic syndromes or cognitive impairment.

B. Assessment of brain structures and volume testing of selected brain structures.

C. Cognitive and functional assessment using clinical tests. All participants groups treated with different RT techniques (three groups) will by randomly divided to two subgroups: exercise subgroup - EG (these are the patients who will have regular cognitive and physical training) and second subgroup (control group - CG).

Analysis of risk in planned study will be connected with failure to reach targeted number of patients (the investigators will enlarge the recruitment pool across additionally cancer hospitals) or increase dropout rate (motivational information will be provided to participants and clinicians). The Greater Poland Cancer Centre has very modern research infrastructure allowing for execution of the proposed project.

Methods of research The study protocol was accepted by the Ethics Committee of Poznan University of Medical Sciences (No. 703/18), and each recruited participant will be given a written informed consent. The investigators will enroll patients with BT using the updated 2016 edition of the World Health Organization Classification of Tumors of CNS which uses molecular parameters and the histology to define the main tumor categories for the first time. The investigators will analyze 150 patients together with three different CNS groups of tumors: from III and IV brain tumor groups, and metastatic tumors. The study will include patients with BT enrolled to RT, between 18-70 y o , in good general health conditions (according to Eastern Cooperative Oncology Group 0-2), after obtaining informed consent for participation in the study. The investigators are planning to exclude patients with numerous tumors (> 2), with psychological or psychiatric illnesses treated pharmacologically, or with other neurological disorders (e.g. sclerosis multiplex, Parkinson's disease, meningitis, etc.), or significant clinical circulatory failure (> III NYHA). Enrolled patients will be treated with the one of three RT techniques in the Department of Radiotherapy: 1) CyberKnife, which relies on precise 3D imaging and localization to deliver ablative doses of radiation to the tumor, and can significantly reduce exposure of healthy brain tissue (18 Gy per dose to total 66 Gy) or 2) IMRT using conventional fractionation of 1.8 Gy per day to total dose 54 Gy or 2 Gy per dose to the total dose 60 Gy) or 3) WBRT as the treatment choice for metastatic tumors - the fractionation schedule used is 30 Gy delivered in 10 fractions or 20 Gy in 5 days. Participants randomly selected to EG will perform cognitive and physical training (120 min./5 times per week during study observation) conducted by rehabilitation staff who will be employed for this project: physiotherapist and neuropsychologist. For neuropsychological rehabilitation, the investigators will use the RehaCom system - a special neurocognitive programs and software. During RT, EG will do physical training (such as cycling, running on properly calibrated equipment as well as neuromuscular reeducation exercises using advanced technical tool - Neuroforma computer software) with maximum heart rate to 70%HRmax. After RT, participants in EG will do special exercise training at home under supervision of the hospital staff. Participants from CG will be provided with normal hospital care during RT and next will conduct a normal daily activity at home. According to the study evaluation plan, all participants will be observed before and after end of RT, and during control visits (T2, T3) at cancer center. Patients' blood samples will be collected in the Laboratory Ward in the morning, before breakfast according to the study plan. The investigators will evaluate individual markers in the Department of Radiobiology in collaboration from the Department of Neurochemistry and Neuropathology at Poznan University of Medical Sciences, because the Radiobiology Laboratory is fully equipped with all specialized, high-tech instruments required for the execution of this project.. In the Department of Rehabilitation in cancer center, all study participants will be evaluated in terms of cognitive and physical functioning. Raw cognitive test scores will be compared with published normative values according to age and to education. The investigators will include in the study evaluation with the use of Mini-Mental State Examination (MMSE), Benton Visual Retention Test (BVRT), California Verbal Learning Test (CVLT), Color trials test (CTT), Wisconsin Card Sorting Test (WCST), Trail Making Test A and B (TMT A & B), Montreal Cognitive Assessment (MoCA) 7.2 scale, and Addenbrooke's Cognitive Examination III (ACE III) test as well as the Psychology Experiment Building Language (PEBL) software for objective evaluation of selected cognitive and behavior functions. For general assessment of physical, psychological and social function the investigators will use the Functional Independence Measures (FIM) scale. This will be an unprecedented study yielding unique results on neuroscience in the process of cancer treatment with modern techniques.

ELIGIBILITY:
Inclusion criteria:

* Patients with three different CNS groups of tumors: from III and IV brain tumor groups, and metastatic tumors enrolled to RT,
* Age between 18-70 years,
* good general health conditions (according to Eastern Cooperative Oncology Group (ECOG) 0-2),
* obtaining informed consent for participation in the study.

Exclusion criteria:

* Patients with numerous tumors (above two),
* psychological or psychiatric illnesses treated pharmacologically,
* neurological disorders (e.g. MS, Parkinson's disease, meningitis, etc.),
* significant clinical circulatory failure (above III NYHA).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Markers of BBB disruption | up to 48 months
  The astrocytic protein S-100β will be estimated using enzyme-linked immunoassay (ELISA).
Circulating tight junction-related proteins | up to 48 months
  To estimate circulating tight junction-related proteins (OCLN, CLDN5, ZO-1) concentrations, rabbit anti - human OCLN antibodies will be used.
Onkoneural antibodies in blood | up to 48 months
  Onconeural antibodies will be identified with indirect immunofluorescence and confirmed with Line blott with the use of recombinants.

SECONDARY OUTCOMES:
Anti-neural antibodies in blood | up to 48 months
  Anti-neural antibodies will be tested by means of indirect immunofluorescence only.
Superficial anti-neuronal antibodies in blood | up to 48 months
  Superficial anti-neuronal antibodies will be identified in patients' serum by means of cell-based assay.
MRI scans and the selected structures of the brain | up to 48 months
  The investigators will assess volumetry and morphology of selected brain structures from MRI scans. Hippocampus, thalamus, cerebellum, brainstem, frontal and tempo-parietal lobes, and total brain volume will be determined from the T1-weighted MRI with FreeSurfer, an automated segmentation tool.

OTHER OUTCOMES:
Neuropsychological Assessment | up to 48 months
  The study will include neurological examination and clinimetric evaluation according the Polish Psychological Association with the use of Montreal Cognitive Assessment (MoCA) 7.2 scale as well as the Psychology Experiment Building Language (PEBL) software for objective evaluation of selected cognitive and behavior functions.
Functional Assessment | up to 48 months
  For general assessment of physical, psychological and social function the investigators will use the Functional Independence Measures (FIM; min. 0 - max.126) system. Higher scores means better outcome. It is the scoring system that may be able to objectively determine impairments in different domains.

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Hojan, MD, PhD, Principal Investigator — Greater Poland Cancer Centre
Locations (1):
- Greater Poland Cancer Centre, Poznan, Greater Poland Voivodeship, Poland

REFERENCES:
- [Background] Attia A, Page BR, Lesser GJ, Chan M. Treatment of radiation-induced cognitive decline. Curr Treat Options Oncol. 2014 Dec;15(4):539-50. doi: 10.1007/s11864-014-0307-3. PMID 25228143
- [Background] Baillieux H, De Smet HJ, Paquier PF, De Deyn PP, Marien P. Cerebellar neurocognition: insights into the bottom of the brain. Clin Neurol Neurosurg. 2008 Sep;110(8):763-73. doi: 10.1016/j.clineuro.2008.05.013. Epub 2008 Jul 7. PMID 18602745
- [Background] Benraiss A, Chmielnicki E, Lerner K, Roh D, Goldman SA. Adenoviral brain-derived neurotrophic factor induces both neostriatal and olfactory neuronal recruitment from endogenous progenitor cells in the adult forebrain. J Neurosci. 2001 Sep 1;21(17):6718-31. doi: 10.1523/JNEUROSCI.21-17-06718.2001. PMID 11517261
- [Background] Blyth BJ, Farhavar A, Gee C, Hawthorn B, He H, Nayak A, Stocklein V, Bazarian JJ. Validation of serum markers for blood-brain barrier disruption in traumatic brain injury. J Neurotrauma. 2009 Sep;26(9):1497-1507. doi: 10.1089/neu.2008.0738. PMID 19257803
- [Background] Fischl B. FreeSurfer. Neuroimage. 2012 Aug 15;62(2):774-81. doi: 10.1016/j.neuroimage.2012.01.021. Epub 2012 Jan 10. PMID 22248573
- [Background] Greene-Schloesser D, Moore E, Robbins ME. Molecular pathways: radiation-induced cognitive impairment. Clin Cancer Res. 2013 May 1;19(9):2294-300. doi: 10.1158/1078-0432.CCR-11-2903. Epub 2013 Feb 6. PMID 23388505
- [Background] Hipkiss AR, Cartwright SP, Bromley C, Gross SR, Bill RM. Carnosine: can understanding its actions on energy metabolism and protein homeostasis inform its therapeutic potential? Chem Cent J. 2013 Feb 25;7(1):38. doi: 10.1186/1752-153X-7-38. PMID 23442334
- [Background] Kanner AA, Marchi N, Fazio V, Mayberg MR, Koltz MT, Siomin V, Stevens GH, Masaryk T, Aumayr B, Vogelbaum MA, Barnett GH, Janigro D. Serum S100beta: a noninvasive marker of blood-brain barrier function and brain lesions. Cancer. 2003 Jun 1;97(11):2806-13. doi: 10.1002/cncr.11409. PMID 12767094
- [Background] Louis DN, et al. (2016) WHO classification of tumours of the central nervous system, ed 4 Lyon, IARC Press
- [Background] Manda K, Ueno M, Anzai K. Cranial irradiation-induced inhibition of neurogenesis in hippocampal dentate gyrus of adult mice: attenuation by melatonin pretreatment. J Pineal Res. 2009 Jan;46(1):71-8. doi: 10.1111/j.1600-079X.2008.00632.x. Epub 2008 Sep 16. PMID 18798786
- [Background] McDuff SG, Taich ZJ, Lawson JD, Sanghvi P, Wong ET, Barker FG 2nd, Hochberg FH, Loeffler JS, Warnke PC, Murphy KT, Mundt AJ, Carter BS, McDonald CR, Chen CC. Neurocognitive assessment following whole brain radiation therapy and radiosurgery for patients with cerebral metastases. J Neurol Neurosurg Psychiatry. 2013 Dec;84(12):1384-91. doi: 10.1136/jnnp-2013-305166. Epub 2013 May 28. PMID 23715918
- [Background] Ming GL, Song H. Adult neurogenesis in the mammalian brain: significant answers and significant questions. Neuron. 2011 May 26;70(4):687-702. doi: 10.1016/j.neuron.2011.05.001. PMID 21609825
- [Background] Mizumatsu S, Monje ML, Morhardt DR, Rola R, Palmer TD, Fike JR. Extreme sensitivity of adult neurogenesis to low doses of X-irradiation. Cancer Res. 2003 Jul 15;63(14):4021-7. PMID 12874001
- [Background] Schulzke JD, Fromm M. Tight junctions: molecular structure meets function. Ann N Y Acad Sci. 2009 May;1165:1-6. doi: 10.1111/j.1749-6632.2009.04925.x. PMID 19538280
- [Background] Sun YX, Chu GL (2010) Expression changes of tight junction proteins ZO-1 and occludin after hypoxic-ischemic brain damage in neonatal rats. Zhongguo Xiandai Yixue Zazhi. 20(21):3210-3213
- [Background] Wen PY, Chang SM, Van den Bent MJ, Vogelbaum MA, Macdonald DR, Lee EQ. Response Assessment in Neuro-Oncology Clinical Trials. J Clin Oncol. 2017 Jul 20;35(21):2439-2449. doi: 10.1200/JCO.2017.72.7511. Epub 2017 Jun 22. PMID 28640707
- [Background] Wu PH, Coultrap S, Pinnix C, Davies KD, Tailor R, Ang KK, Browning MD, Grosshans DR. Radiation induces acute alterations in neuronal function. PLoS One. 2012;7(5):e37677. doi: 10.1371/journal.pone.0037677. Epub 2012 May 25. PMID 22662188
- [Background] Voss MW, Prakash RS, Erickson KI, Basak C, Chaddock L, Kim JS, Alves H, Heo S, Szabo AN, White SM, Wojcicki TR, Mailey EL, Gothe N, Olson EA, McAuley E, Kramer AF. Plasticity of brain networks in a randomized intervention trial of exercise training in older adults. Front Aging Neurosci. 2010 Aug 26;2:32. doi: 10.3389/fnagi.2010.00032. eCollection 2010. PMID 20890449